CLINICAL TRIAL: NCT06629844
Title: Education Program for Enhancing Attitude Toward People Living With Dementia Among Healthcare Students Using Virtual Reality: Pilot Study
Brief Title: Enhancing Healthcare Students' Attitudes Toward Dementia Care Through Virtual Reality Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Airlangga (Other)
Collaborators: Tokyo University (Other)
Responsible Party: Principal Investigator, Dianis Wulan Sari, Principal Investigator, Universitas Airlangga
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3359-KEPK; 23KK0168 (Other Grant/Funding Number: Japan Society for the Promotion of Science)
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Nursing Students; Education Program on Dementia
Keywords: Aged; Dementia; Education Program; Healthcare Student; Long-term care; Virtual Reality
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Program (Experimental): The experiment group will receive the VR dementia education program, which will be conducted once for each participant.
  Interventions: Other: The VR dementia education group
- Standard Course Material (Active Comparator): The control group will receive the standard course material through the university's e-learning platform.
  Interventions: Other: The control group

INTERVENTIONS:
Other: The VR dementia education group — The intervention group will receive the VR dementia education program, which will be conducted once for each participant, and each session will accommodate a maximum of 20 participants. The VR dementia education program will follow the flow below, integrating video dramatizations, VR experiences, lectures, and discussions. The program is designed to simulate real-life dementia care situations, encourage reflection, and enhance nursing students' understanding of dementia management. The following are the steps for intervention: Introduction (3 minutes), Pre-Program Questionnaire (10 minutes), Lecture Introduction (2 minutes), Bad Drama (Unfriendly Communication) (10 minutes), Bad VR (10 minutes), Discussion (5 minutes), Lecture 1: What is Dementia? (10 minutes), Good VR (10 minutes), Good Drama (10 minutes), Lecture 2: What Can We Do to Support PLWD? (5 minutes), N-impro (10 minutes), Post-Program Questionnaire (10 minutes), Conclusion (5 minutes).
  Arms: Virtual Reality Program
Other: The control group — The intervention begins with an introduction to the VR dementia program, outlining its objectives and setting participant expectations. A pre-program questionnaire follows to assess baseline knowledge, attitudes, and intention to assist people with dementia. A brief lecture introduces a dramatization showing ineffective communication with a PLWD, followed by a VR scenario highlighting poor care practices. After discussing these observations, participants attend a lecture explaining dementia's symptoms and progression, with culturally adapted video content for Indonesian audiences. Next, a positive VR scenario demonstrates best practices in dementia care, followed by a video on supportive communication. A second lecture offers practical strategies for caregiving and communication, complemented by an N-impro session to deepen understanding. The session concludes with a post-program questionnaire and final reflection to encourage real-world application of the learned skills.
  Arms: Standard Course Material

SUMMARY:
This quasi-experimental study focuses on Indonesian nursing students and aims to examine the effectiveness of virtual reality (VR) dementia educational programs. The study addresses the following research questions:

1. What is the current state of knowledge and awareness about dementia among participants before engaging in a VR dementia education program?
2. What is the effect of a VR dementia education program on improving participants' attitude, knowledge, and intention to help toward people living with dementia, and how are participants satisfied with the VR dementia education program? Participants will voluntarily join a 120-minute class education program, with each participant attending only once. The program, integrated into the faculty's dementia-related courses, will be structured around a series of components, including introduction, pre-program questionnaire, lecture, bad drama (unfriendly communication), bad version of VR, discussion, Lecture (about dementia), good VR, good drama, Lecture, N-impro, post-program questionnaire, and conclusion.

The VR education program will be included in dementia-related courses in the faculty of nursing.

DETAILED DESCRIPTION:
This quasi-experimental study aims to evaluate a virtual reality (VR) dementia education program among nursing students in Indonesia. The participants will be nursing students who are enrolled in specific semesters and courses designated for the implementation of this educational program. At Universitas Airlangga, the study will be conducted with students in the fifth semester (third year). All prospective participants will be assigned new ID numbers to ensure the confidentiality of their student ID numbers. This protocol has been reviewed and approved by the Faculty of Nursing's Ethics Committee at Universitas Airlangga.

The VR dementia education program will be integrated into the Psychiatric Nursing class, which covers themes related to dementia care. Participants will be recruited during the Psychiatric Nursing course through class announcements. An overview of the research process will be provided, and detailed instructions regarding the study will be given shortly before it begins. The research team will announce the study approximately one week in advance, and recruitment will occur via Google Forms. Selected participants will receive their new ID numbers and details about the program's schedule and location through a class announcement three days before the intervention.

On the day of the intervention, participants will attend the designated location and sign an attendance sheet using their new IDs. The Principal Investigator (PI) will explain the study's stages and emphasize that participants can withdraw at any time without any consequences. Participation in the study will be entirely voluntary, and there will be no coercion. Students who opt out of the study will still receive standard dementia-related material through the university's e-learning platform. Still, they will not participate in the game-based education program. Students who agree to participate in the study will provide informed consent. Those in the program will complete a questionnaire before and after the intervention.

Regarding recruitment, eligible participants will be identified through the university's e-learning portal. Students registered in the selected courses for the 2024/2025 academic year will be noted at the beginning of the semester. All eligible students will receive comprehensive information about the study and an invitation to participate.

The research team will explain the program in person and provide written explanations at the start of the Psychiatric Nursing course. The 2024/2025 Psychiatric Nursing course consists of four classes, each with 50-60 students. One class will be randomly selected to participate in this pilot study as the intervention group. The remaining three classes will serve as the control group, receiving standard course material through the e-learning platform. Both the intervention and control groups will complete pre- and post-intervention questionnaires. Data will be collected again from both groups at the end of the Psychiatric Nursing course (expected in January 2025) to measure the long-term effects.

The intervention group will receive the VR dementia education program, while the control group will attend a standard lecture. Both interventions will be conducted once. The control group will receive a single lecture via the e-learning platform. Students who provide informed consent will be asked to complete the baseline survey (T1). In the intervention group, students will attend a classroom lecture and discussion on dementia (1st class) and then complete a post-lecture survey (T2). Later, they will be asked to complete another post-lecture survey (T3) at the end of the semester. The control group will follow the same timeline for completing the surveys (T1-T3).

ELIGIBILITY:
Inclusion Criteria:

- Nursing students enrolled in the designated semester and courses that align with the program's implementation at Universitas Airlangga.

Exclusion Criteria:

- Students who are not enrolled in the specified semester and courses or those who have prior experience with similar VR dementia education programs could influence the results.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Attitudes Toward People with Dementia Scale | 3-5 minutes for completion of the questionnaire
  Participants' attitudes toward persons living with dementia (PLWD) will be assessed using the Attitudes Toward People with Dementia Scale. Factors related to attitudes toward people with dementia: Development of the Attitude Toward Dementia Scale and Dementia Knowledge Scale. The original scale was published in Japanese, and a forward-backward translation process was conducted to produce the Indonesian version of the scale.
  The questionnaire consists of 14 items and it is designed to evaluate participants' attitudes toward PLWD. The total score ranged from 14 to 56, with high scores indicating favorable attitudes.

SECONDARY OUTCOMES:
Knowledge of Dementia | 3-5 minutes for completion of the questionnaire
  Participants' knowledge of dementia will be assessed using the Dementia Knowledge Scale. This scale was originally designed to measure various aspects of dementia knowledge, including symptoms, causes, progression, and caregiving strategies. The scale consists of 15 multiple-choice and true/false questions that cover a broad range of dementia-related topics. The Indonesian version of the scale was created through a forward-backward translation process to ensure cultural and linguistic accuracy. This scale will require respondents to provide answers using a 3-point Likert scale ranging from agree, disagree, and don't know. The author will calculate the total dementia knowledge score, with a high score indicating a high level of knowledge about dementia.
Intention to Help Persons Living with Dementia (PLWD) | 2-3 minutes for completion of the vignettes
  To assess participants' intention to help PLWD, we will use a set of four vignettes based on the previous study. Each vignette presents a realistic scenario in which a person with dementia may need assistance, such as confusion in a public place, difficulty with daily tasks, or issues related to memory loss. Participants will read through each vignette and indicate their intended helping behavior on a 4-point Likert scale (ranging from "definitely would not help" to "definitely would help"). The vignettes are designed to assess the participants' willingness to offer practical, emotional, or social support to PLWD in everyday situations. The Indonesian version of the vignettes and Likert scale has also undergone a forward-backward translation to ensure that the language and context are appropriate for Indonesian nursing students. A high score indicates a high intention to help people living with dementia.
User Experience Questionnaire (UEQ) | 3-5 minutes for completion of the questionnaire
  To assess participants' perceptions of the VR dementia education program, we will use the User Experience Questionnaire (UEQ). This questionnaire evaluates users' experiences with the VR program across several dimensions, such as attractiveness, perspicuity, efficiency, dependability, stimulation, and novelty. The UEQ was used previously in similar studies and provided valuable feedback on the user experience. The Indonesian version of the UEQ https://www.ueq-online.org/, will be employed to ensure the questionnaire is culturally and linguistically appropriate. It typically involves a series of semantic differential scales, and the responses are scored from -3 to +3. Higher scores indicate a more positive perception of the user experience.

CONTACTS AND LOCATIONS:
Overall Officials: Dianis Wulan Sari, Ph.D, Principal Investigator — Faculty of Nursing, Universitas Airlangga
Locations (1):
- Faculty of Nursing, Universitas Airlangga, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
The IPD associated with participants'; real IDs will be retained only by the PI of this study.
  New datasets will use new IDs so that only the PI can link the research data to participants' original IDs.
  Datasets that use the new IDs will be shared with the research team for data processing purposes (statistical analysis plan, SAP) and publication. All data will be stored for five years (Oktober 2024-Oktober 2029).
  Datasets will not be made public and will only be shared with the project's research team.

REFERENCES:
- [Background] Sari DW, Igarashi A, Takaoka M, Yamahana R, Noguchi-Watanabe M, Teramoto C, Yamamoto-Mitani N. Virtual reality program to develop dementia-friendly communities in Japan. Australas J Ageing. 2020 Sep;39(3):e352-e359. doi: 10.1111/ajag.12797. Epub 2020 Jun 2. PMID 32483931
- [Background] Wu J, Igarashi A, Suzuki H, Matsumoto H, Kugai H, Takaoka M, Yamamoto-Mitani N. Effects of a dementia educational programme using virtual reality on nurses in an acute care hospital: A pre-post comparative study. Int J Older People Nurs. 2024 May;19(3):e12616. doi: 10.1111/opn.12616. PMID 38769648
- [Background] Suzuki H, Igarashi A, Matsumoto H, Kugai H, Takaoka M, Sakka M, Ito K, Hagiwara Y, Yamamoto-Mitani N. A Dementia-Friendly Educational Program Using Virtual Reality for the General Public in Japan: A Randomized Controlled Trial for DRIVE. Gerontologist. 2024 Nov 1;64(11):gnae113. doi: 10.1093/geront/gnae113. PMID 39140623
- [Background] Igarashi A, Matsumoto H, Takaoka M, Kugai H, Suzuki M, Yamamoto-Mitani N. Educational Program for Promoting Collaboration Between Community Care Professionals and Convenience Stores. J Appl Gerontol. 2020 Jul;39(7):760-769. doi: 10.1177/0733464819871878. Epub 2019 Sep 3. PMID 31478434
- [Background] Matsumoto H, Hagiwara Y, Yamamoto-Mitani N, Igarashi A. A Randomized Control Trial for ReDeSign: A Dementia-Friendly Mobile Microlearning Training for Store Workers in Japan. Gerontologist. 2023 Sep 2;63(8):1300-1310. doi: 10.1093/geront/gnac182. PMID 36508394
- [Background] GBD 2021 Demographics Collaborators. Global age-sex-specific mortality, life expectancy, and population estimates in 204 countries and territories and 811 subnational locations, 1950-2021, and the impact of the COVID-19 pandemic: a comprehensive demographic analysis for the Global Burden of Disease Study 2021. Lancet. 2024 May 18;403(10440):1989-2056. doi: 10.1016/S0140-6736(24)00476-8. Epub 2024 Mar 11. PMID 38484753
- [Background] Leroi I, Kitagawa K, Vatter S, Sugihara T. Dementia in 'super-aged' Japan: challenges and solutions. Neurodegener Dis Manag. 2018 Aug;8(4):257-266. doi: 10.2217/nmt-2018-0007. Epub 2018 Jul 24. PMID 30040019
- [Background] Igarashi A, Eltaybani S, Takaoka M, Noguchi-Watanabe M, Yamamoto-Mitani N. Quality Assurance in Long-Term Care and Development of Quality Indicators in Japan. Gerontol Geriatr Med. 2020 Nov 27;6:2333721420975320. doi: 10.1177/2333721420975320. eCollection 2020 Jan-Dec. PMID 35047653
- [Background] Matsumoto H, Igarashi A, Suzuki M, Yamamoto-Mitani N. Association between neighbourhood convenience stores and independent living in older people in Japan. Australas J Ageing. 2019 Jun;38(2):116-123. doi: 10.1111/ajag.12607. Epub 2019 Jan 30. PMID 30701659